CLINICAL TRIAL: NCT05593666
Title: A Phase II, Multicentre, Randomized, Two-arm Blinded Study to Assess the Efficacy and Safety of Two LXE408 Regimens for Treatment of Patients With Primary Visceral Leishmaniasis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DNDi-LXE408-01-VL; CLXE408A12201R (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Primary Visceral Leishmaniasis
MeSH Terms: interventions — LXE408; liposomal amphotericin B

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LXE408 short regimen (Experimental): LXE408 once daily for seven days (followed by 7 days of placebo).
  Interventions: Drug: LXE408; Other: Placebo
- LXE408 long regimen (Experimental): LXE408 once daily for 14 days
  Interventions: Drug: LXE408
- Standard of care (Active Comparator): AmBisome® 10 mg/kg IV single dose (SDA)
  Interventions: Drug: AmBisome®

INTERVENTIONS:
Drug: LXE408 — Film-coated tablets
  Arms: LXE408 long regimen; LXE408 short regimen
Other: Placebo — Placebo film-coated tablets
  Arms: LXE408 short regimen
Drug: AmBisome® — Sterile lyophilised powder in a 15 mL sterile clear glass vial
  Arms: Standard of care

SUMMARY:
This is a phase II, multicentre, randomized, two-arm blinded study with an open label calibrator arm in adults and adolescents (≥12 years) with confirmed primary VL.

DETAILED DESCRIPTION:
This study is run by DNDi with Novartis as co-development partner

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years (at the time of the screening visit) who are able to comply with the study protocol. Following a favourable interim analysis result, patients ≥12 <18 years will also be enrolled in the trial
* Patients for whom written informed consent has been obtained (if aged 18 years and over) or signed by parent(s) or legal guardian for patients under 18 years of age. In the case of minors, assent from the child also needs to be obtained
* Primary symptomatic VL (defined as typical parameters including, but not limited to, fever for > 2 weeks, weight loss, and splenomegaly)
* Visualization of Leishmania amastigotes by microscopy in tissue samples (spleen or bone marrow)

Exclusion Criteria:

* Clinical signs of severe VL (jaundice, spontaneous bleeding, edema, ascites, coma, organ failure)
* Laboratory abnormalities including ALT/SGPT > 3 times ULN, total bilirubin > 1.5 times ULN, creatinine >1.5 times ULN, amylase or lipase > 1.5 times ULN, haemoglobin < 6 g/dL or other clinically significant abnormal laboratory parameters which, in the opinion of the investigator, may indicate severe VL
* Patients with history of previous leishmaniasis and confirmed relapse
* Patients with para-kala-azar dermal leishmaniasis
* Patients with severe malnutrition (for children ≥12-<18 years: BMI-for-age WHO reference curves by sex, z score < -3; for adults ≥18 years: BMI < 16)
* History of congenital or acquired immunodeficiency, including positive HIV (test at screening)
* Known hypersensitivity to amphotericin B deoxycholate or any other constituents of AmBisome®
* Concomitant infections such as tuberculosis, severe malaria, or any other serious underlying disease that may interfere with the disease assessment (e.g., cardiac, renal, hepatic, haematologic, and pancreatic)
* Infection with hepatitis B (HBV) or hepatitis C virus (HCV). A positive HBV surface antigen (HBsAg) test, or if standard local practice, a positive HBV core antigen test, excludes a subject. Patients with a positive HCV antibody test should have HCV RNA levels measured. Patients with positive (detectable) HCV RNA should be excluded.
* Pregnant or nursing (lactating) women
* Women of childbearing potential who do not accept to have a pregnancy test done at screening and/or who do not agree to use highly effective contraception while taking the investigational drug and for 5 half-lives or 5 days, whichever is longer, after stopping the investigational drug.
* Sexually active males unwilling to use a condom during intercourse while taking the investigational drug and for 5 half-lives or 5 days, whichever is longer, after stopping the investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with initial cure at Day 28 for LXE408 | Day 28
  Initial cure defined as clinical improvement of Visceral leishmaniasis (VL), absence of parasites in the spleen or bone marrow (microscopy), and no rescue therapy on or before Day 28.

SECONDARY OUTCOMES:
Proportion of patients with initial cure at Day 28 for AmBisome® | Day 28
  Initial cure defined as clinical improvement of Visceral leishmaniasis (VL), absence of parasites in the spleen or bone marrow (microscopy), and no rescue therapy on or before Day 28.
Proportion of patients with definitive cure at Day 180 for LXE408 and AmBisome® | Day 180
  Definitive cure described as initial cure at Day 28, no requirement for rescue treatment throughout the study, no death associated to VL and absence of any clinical parameters of VL at Day 180.
Mortality | Days 28 and 180
  All-cause mortality and mortality not associated with Visceral leishmaniasis (VL)
Cmax for LXE408 | Days 1 and 7
  Maximum Observed Blood-drug Concentrations for LXE408
Tmax for LXE408 | Days 1 and 7
  Time to Reach Maximum Blood-drug Concentrations for LXE408
AUCtau for LXE408 | Days 1 and 7
  Area Under The Plasma Concentration-time Curve Over A Dosing Interval for LXE408
CLss/F for LXE408 | Days 1 and 7
  Apparent Clearance for LXE408
Cmax for Amphotericin B | Days 1 and 7
  Maximum Observed Blood-drug Concentrations for Amphotericin B
AUC0-24h for Amphotericin B | Day 1
  Area under the plasma concentration-time curve from time zero to 24h for Amphotericin B
AUC0-infinity for Amphotericin B | Day 1
  Area under the plasma concentration-time curve from time zero to infinity for Amphotericin B
Blood parasite clearance | Baseline and Days 1, 3, 5, 7, 10, 14, 28 and 56
  Blood parasite clearance over time, as measured by quantitative polymerase chain reaction (qPCR) from blood samples at defined time points and at any suspicion of relapse during the trial.
Proportion of patients with a positive loop-mediated isothermal amplification (LAMP) from blood samples | Baseline and Days 28 and 56
  Proportion of patients with a positive loop-mediated isothermal amplification (LAMP) from blood samples at defined time points and at any suspicion of relapse during the trial.
Tissue parasite loads | Baseline and Day 28
  Tissue parasite loads, as measured by qPCR from tissue samples (spleen or bone marrow) collected at defined time points and at any suspicion of relapse during the trial.
Proportion of patients with a positive loop-mediated isothermal amplification (LAMP) from tissue samples | Baseline and Day 28
  Proportion of patients with a positive loop-mediated isothermal amplification (LAMP) from tissue samples at defined time points and at any suspicion of relapse during the trial.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - DrugsNeglectedD Investigational Site, Bihār
  - DrugsNeglectedD Investigational Site, Patna

IPD SHARING:
Plan to Share IPD: Undecided